CLINICAL TRIAL: NCT01202097
Title: A PHASE III, RANDOMIZED, OPEN-LABEL, NON-INFERIORITY COMPARATIVE STUDY BETWEEN SERETIDE® 50/250 ΜG and SALMETEROL/FLUTICASONE SINGLE INHALATION CAPSULE 50/250 ΜG EUROFARMA in PATIENTS with ASTHMA
Brief Title: A Non- Inferiority Comparative Study Between Seretide® and Salmeterol/Fluticasone Eurofarma in Patients with Asthma
Acronym: CAINAS SF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF113
Record Dates: First submitted 2010-09-14; First posted 2010-09-15 (Estimated); Last update posted 2025-03-31 (Actual); Status verified 2010-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Salmeterol/Fluticasone (Experimental)
  Interventions: Drug: Salmeterol/Fluticasone
- Seretide (Active Comparator)
  Interventions: Drug: Seretide

INTERVENTIONS:
Drug: Salmeterol/Fluticasone
  Arms: Salmeterol/Fluticasone
Drug: Seretide
  Arms: Seretide

SUMMARY:
The primary objective will be to compare the formulations regarding their impact on the pulmonary function of persistent asthma patients and the secondary objective will be the clinical control of the disease's symptoms.

DETAILED DESCRIPTION:
The primary objective will be to compare the formulations regarding their impact on the pulmonary function of persistent asthma patients and the secondary objective will be the clinical control of the disease's symptoms.

Primary endpoint: Forced expiratory volume in 1 second (FEV1) at the final visit.

Secondary endpoints: Expiratory Flow Peak (EFP), symptoms score, FEV1 throughout the study, use of rescue medication, compliance with inhaler use, inhaler acceptance and preference, and frequency of the observed adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Sign the ICF
* ≥ 12 years old
* Have a persistent asthma diagnosis, as per GINA classification,18 with symptoms for at least 6 months and clinically stable for at least 1 month with the ACQ-7 test (please see Appendix C) ≤ 3.0
* Current use of inhaled corticosteroid (up to 1000 µg of beclomethasone dipropionate) whether combined or not with long-term β2-adrenergics and relief medication (salbutamol or equivalent)
* Initial FEV1 of at least 40% of the normal value expected
* Blood cortisol evaluation within the normal limits.

Exclusion Criteria:

* Use of oral or parenteral corticosteroid within the last 3 previous months to the study
* Hospitalization needed due to asthma within the last 3 previous months to the study
* Active smokers, defined as the consumption of cigarettes, pipes, cigars or any other form of smoking in any amount within the last 3 months
* Presence of severe co-morbidities, such as cardiovascular, renal, liver, neurological, neoplastic, hematological, infectious, dermatological, neurological or psychiatric disease or chronic respiratory disease other than asthma
* Recent (<6 months) or expected participation during this study in other clinical trials involving drugs of any nature or in studies consisting of any - Intolerance or allergy to any component of the drugs evaluated in the study
* Pregnant or lactating women
* Chronic use of routine β-blockers, orally or intravenously, including ophthalmic solutions.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2011-08; Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) at the final visit.

SECONDARY OUTCOMES:
Expiratory Flow Peak (EFP)

CONTACTS AND LOCATIONS:
Locations (6):
- Brazil (6):
  - Hospital de Clinicas UFPR, Curitiba, PR
  - Centro de Referencia em Enfermidades Respiratoria e Alergica, Salvador, BA
  - Centro de Estudos de Pneumologia FMABC, São Paulo
  - IMA Brasil - Instituto de Pesquisa Clínica e Medicina Avançada, São Paulo
  - Stelmach Pesquisa Clinica, São Paulo
  - Clinica de Alergia Martti Antila, Sorocaba, SP